CLINICAL TRIAL: NCT02922283
Title: [18F]FB-IL2 Imaging of T Cell Response as Biomarker to Guide Treatment Decisions in Metastatic Melanoma Patients
Brief Title: IL2 Imaging in Metastatic Melanoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After an interim analysis of the data, it became clear that the imaging results did not correlate to the primary outcome measures in this subset of patients.
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22102014
Record Dates: First submitted 2015-12-14; First posted 2016-10-04 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma
Keywords: T cell response; Interleukin 2; PET scan; Ipilimumab; Pembrolizumab; Nivolumab
MeSH Terms: conditions — Melanoma | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IL2-PET scan (Experimental): [18F]FB-IL2 PET scan, Tumor biopsy, CT scan, Biopsy of non-target tissue
  Interventions: Device: IL2-PET scan; Procedure: Tumor biopsy; Device: CT scan; Procedure: Biopsy of non-target tissue

INTERVENTIONS:
Device: IL2-PET scan — All patients in this study will undergo a IL2 PET scan at baseline and week 6 of treatment with immunotherapy.
  Other Names: [18F]FB-IL2 PET scan
Procedure: Tumor biopsy — A procedure to acquire tissue of a predetermined melanoma metastasis will be performed in all patients that participate in phase 2 of this study.
Device: CT scan — A CT scan of diagnostic quality will accompany all the PET scans and will additionally been made 12 and 16 weeks after start of immunotherapy to evaluate response to treatment.
Procedure: Biopsy of non-target tissue — A biopsy of skin and colon non-target tissue involved in an immune-related side effect is optional in patients that participate in phase 2 of this study.

SUMMARY:
T cell infiltration of tumor lesions is a known prognostic factor in several tumor types and is used as treatment mechanism in some of these tumor types. In metastatic melanoma, treatment with immune checkpoint inhibitors induces clinical benefit in about 30-50% of the patients. These immune-based therapies are however accompanied by serious immune-related adverse events and high costs.

Tumor infiltrating T cells express the high affinity interleukin-2 (IL2) receptor on their surface. These T cells could therefore be visualized by molecular imaging with a radio-labelled ligand for this receptor. For this purpose, the investigators have developed the PET tracer [18F]FB-IL2.

The study commences with a biodistribution study (phase 1) in 5 subjects. Thereafter the main study (phase 2) starts, in which 25 subjects will receive two [18F]FB-IL2 PET scans at baseline and week 6 of treatment with either ipilimumab, nivolumab, pembrolizumab or the combination of ipilimumab and nivolumab. If [18F]FB-IL2 PET is able to detect a response to treatment, it could serve as a non-invasive early indicator of T cell response to the treatment. Besides, accumulation of the PET tracer in non-target tissue could indicate infiltration of activated T cells in normal organs and thus may predict the development of an immune-related adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed informed consent.
2. ≥18 years of age.
3. Histologically confirmed cutaneous metastatic melanoma (Stage IV).
4. Evidence of at least one measurable metastatic lesion based on RECIST version 1.1.
5. At least one easy accessible metastatic melanoma lesion, of which biopsy can be performed.
6. Eligible for treatment with ipilimumab, nivolumab, pembrolizumab, or the combination of ipilimumab and nivolumab.
7. No contraindication for performing a CT scan.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
9. Women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study.
10. Must have adequate organ function (e.g. liver, kidney) as defined

Exclusion Criteria:

1. Pre-existing auto-immune disease, which could be exacerbated by ipilimumab (e.g. Crohn, Hashimoto's Thyroiditis).
2. Presence of malignancy other than the disease under study within 5 years of study enrolment. Subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
3. Brain metastases that are symptomatic or not stable for 8 weeks (must be documented by imaging).
4. The use of corticosteroids (at the start of treatment). Note: Corticosteroids are allowed during the study for immune-related toxicity of immunotherapy, as this will not interfere with activity of immunotherapy.
5. Evidence of active infection requiring antibiotic therapy at start of treatment.
6. Current use of a prohibited medication or requirement of any of these medications during treatment with immune-checkpoint inhibitors as mentioned in the summary of product characteristics (SPC) for Yervoy, Opdivo, and Keytruda.
7. Known immediate or delayed hypersensitivity reaction to ipilimumab, nivolumab or pembrolizumab or excipients.
8. Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0. Grade 2 or higher from previous anti-cancer therapy, except alopecia.
9. A history or evidence of cardiovascular risk including any of the following:

   1. A history or evidence of current clinically significant uncontrolled arrhythmias;
   2. A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization.
   3. A history or evidence of current ≥Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines.
   4. Abnormal cardiac valve morphology (≥grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
   5. Presence of cardiac metastases.
10. Any serious or unstable pre-existing medical conditions (i.e. diabetes mellitus, hypertension, etc), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
11. Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
12. Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Biodistribution and kinetics of [18F]FB-IL2. | 2 hours
  Biodistribution and kinetics will be assessed in the first five patients that participate in this trial (phase 1). A 60-minute dynamic PET scan of the chest and 2 total-body PET scans at 60 and 120 minutes will be acquired to determine tracer kinetics and residence time of the tracer in major organs.
The ability of the [18F]FB-IL2 PET to detect a treatment-induced immune response in tumors. | 6 weeks
  For detection of a treatment-induced immune response the absolute tracer uptake in tumor lesions will be compared between the scan at baseline and the scan after 6 weeks of treatment with ipilimumab, nivolumab, pembrolizumab or the combination of ipilimumab and nivolumab.
Correlation between tumor uptake of [18F]FB-IL2 with the number of IL2 receptor positive immune cells. | 2 days
  The amount of IL2 receptor positive cells will be scored by immunohistochemical staining of tumor biopsy material and will be correlated to the tumor uptake of [18F]FB-IL2.

SECONDARY OUTCOMES:
Correlation between tumor uptake of [18F]FB-IL2 with response to therapy. | 16 weeks
  The increase in tumor uptake of [18F]FB-IL2 ofu the tumor lesions on the PET scan at baseline and week 6 of treatment with immunotherapy, will be correlated to radiological response as measured on the CT scans at week 6, 12 and 16 according to the RECIST 1.1 criteria.
To analyze heterogeneity in immune response to treatment between separate lesions, as determined by [18F]FB-IL2 PET. | 16 weeks
  Both the heterogeneity between separate lesions in one patient and between lesions in different patients will be determined and if possible will be correlated to treatment response (lesion based).
Treatment induced immune cell activation in non-target tissues and if possible the correlation of PET observations with side effects related to the tissue involved. | 16 weeks
  Treatment induced immune cell activation in non-target tissue will be determined by visually comparing the PET results at baseline and after 6 weeks of treatment. In regions with a higher tracer uptake on the week 6 scan the absolute uptake will be determined and this will be correlated to the development of an immune-related adverse event. In case of immune-related side effects localized to the skin or colon, biopsy samples are optional and tissue infiltration of IL2 receptor positive cells can be correlated to [18F]FB-IL2 uptake on PET.
Adverse events of [18F]FB-IL2 PET. | 16 weeks
  Adverse events will be recorded. Vital signs and blood parameters will be determined before and after tracer injection and directly after the PET scan for safety reasons.

CONTACTS AND LOCATIONS:
Overall Officials: G. A. Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van de Donk PP, Wind TT, Hooiveld-Noeken JS, van der Veen EL, Glaudemans AWJM, Diepstra A, Jalving M, de Vries EGE, de Vries EFJ, Hospers GAP. Interleukin-2 PET imaging in patients with metastatic melanoma before and during immune checkpoint inhibitor therapy. Eur J Nucl Med Mol Imaging. 2021 Dec;48(13):4369-4376. doi: 10.1007/s00259-021-05407-y. Epub 2021 Jun 2. PMID 34076745